CLINICAL TRIAL: NCT01111929
Title: Emergency Contraception as a Back up of Lactational Amenorrhea Method of Contraception
Brief Title: Emergency Contraception as a Back up of Lactational Amenorrhea Method(LAM)
Acronym: ECLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mamdouh Shaaban, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECLAM
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy During Breastfeeding; Lactational Amenorrhea Method
Keywords: Emergency contraception; pregnancy during breastfeeding; Lactational amenorrhea Method; unplanned pregnancy
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling for LAM (Active Comparator): Will receive proper postpartum counseling for LAM by trained research nurse. This is in addition to, adequate contraceptive counseling including information about LAM and its prerequisites.
  Women that choose to use LAM will be advised to return to our contraception outpatient clinic to have a long term method of contraception as soon as any of the requirements of LAM expires.
  Interventions: Drug: Counseling for LAM+ LNG-EC
- Counseling for LAM+ LNG-EC (Experimental): LAM counseling and contraceptive counseling +two 0.75 mg Levonorgestrel EC pills
  Interventions: Drug: Counseling for LAM+ LNG-EC

INTERVENTIONS:
Drug: Counseling for LAM+ LNG-EC — They will be provided by the above proper LAM counseling and contraceptive counseling. Additionally, they will be provided by EC pills and advised to use these pills if one of the prerequisites of LAM expires and sexual relation with their husband had occurred before the initiation of another long term contraceptive. Each women in this group will be supplied with one packet containing two 0.75 mg Levonorgestrel EC pills and advised to swallow the two tablets as soon as possible after having sexual intercourse with their husband after the expiry of LAM. They will be informed that they should not use the method after more than 5 days of having intercourse.
  They will be also advised not to use EC pills more than once. All women who have used the EC pills need to visit the clinic within few days of use for contraception advice. All the above information will be additionally given to the patient in a small flyer.

SUMMARY:
Prolonged breast-feeding is an encouraged tradition in Egypt. Breastfeeding is associated with variable degrees of amenorrhea and infertility but there is a risk of resumption of fertility and therefore, of conception during lactation. A consensus statement formalized the lactational amenorrhea method of contraception (LAM), which has subsequently been included in the family planning programs in some developing countries. It has proved to be effective with cumulative pregnancy rates ranging from only 0.9% to 1.2%. However, if any of the prerequisites of LAM expire at any time, the contraceptive efficacy will be much reduced.

The expiry of LAM requirements can occur unexpectedly at a time the woman is not ready to visit a clinic to initiate another contraceptive. Pregnancy during breast-feeding may result in mistimed, unplanned and sometimes unwanted childbirth. A study done in Egypt has shown that one in 4 of pregnancies during lactation were unplanned Such pregnancies, in addition to their negative social impact may lead some women to seek induced abortion; a procedure which, in settings (like Egypt) where abortion is illegal (except on very restricted grounds), is often unsafe.

Levonorgestrel 1.5 mg EC pills has been used for long time and proved to decrease the incidence of pregnancy by 75-85% in each act of unprotected sexual intercourse. Its safety has been documented. It can be used safely during lactation and has been classified by the WHO medical eligibility criteria for contraception as category-1 for lactating mother. Even if take early in pregnancy it is not abortifacient and does not by any mean affect the continuation of pregnancy or cause any side effects to the growing baby (WHO category 1).

The present study tries to estimate the efficacy of in advance provision of 1.5 Levonorgestrel EC pills (as a back-up of LAM) at the time of counseling of LAM when used in increasing the incidence of initiation of another long term method of contraception and probably decreasing the incidence of unintended pregnancy during breast-feeding in rural Egypt.

The investigators are planning to include all women who deliver in the investigators service and intent to breast-feed and planning of birth spacing. Women who refused to participate or planned to use a method of contraception other than LAM and those with expected difficulty of subsequent communication were excluded from participation.

All eligible participants will receive proper counseling for LAM by trained research nurse.

Women who choose to use LAM will be advised to return to the investigators contraception outpatient clinic to have a long term method of contraception as soon as any of the requirements of LAM expires. All eligible participants who accept to participate in the study will be randomly assigned to one of two groups:Group 1 will only receive the above described care (control group). Group II (Intervention group) in which women will have the above proper counseling. Additionally, they will be advised to use the EC pills if one of the prerequisites of LAM expires and sexual relation with their husband had occurred before the initiation of another contraceptive. Each women assigned to the intervention group will be supplied with one packet containing two 0.75 mg Levonorgestrel emergency contraceptive (EC) pills and advised to swallow the two tablets as soon as possible after having sexual intercourse with their husband after the expiry of LAM. They will be informed that they should not use the method after more than 5 days of having intercourse. They will be also advised not to use EC pills more than once. All women who have used the EC pills need to visit the clinic within few days of use for contraception advise. All the above information will be additionally given to the patient in a small flyer.

ELIGIBILITY:
Inclusion Criteria:

* All women who delivers in the obstetric intent to breast-feed.
* Eligible participants should have been planning of birth spacing

Exclusion Criteria:

* Women refusal to participate in the study
* Women planned to use a method of contraception other than LAM
* Anticipation of difficulty of subsequent communication with the woman

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1174 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Initiation of long term contraception with 6 month postpartum | 6 month

SECONDARY OUTCOMES:
Use/non-use of EC pills | 6 months
Use/non-use of any other type of EC ( e.g insert IUD if eligible) | 6 months
Pregnancy rate in each group | 6 months
Side effects of LNG EC pills | 6 months
The prevalence of unwanted pregnancy in each study group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Omar M Shaaban, MD, Principal Investigator — Department of Obstetrics and Gynecology, Assiut University, Egypt

REFERENCES:
- [Background] Shaaban MM, Kennedy KI, Sayed GH, Ghaneimah SA, Abdel-Aleem AM. The recovery of fertility during breast-feeding in Assiut, Egypt. J Biosoc Sci. 1990 Jan;22(1):19-32. doi: 10.1017/s0021932000018344. PMID 2298758
- [Derived] Shaaban OM, Hassen SG, Nour SA, Kames MA, Yones EM. Emergency contraceptive pills as a backup for lactational amenorrhea method (LAM) of contraception: a randomized controlled trial. Contraception. 2013 Mar;87(3):363-9. doi: 10.1016/j.contraception.2012.07.013. Epub 2012 Aug 27. PMID 22935323